CLINICAL TRIAL: NCT06862401
Title: Influence of Sequential Practicing for Psychomotor Skill Acquisition of Non-dominant Hand in Undergraduate Dental Students: A Randomized Controlled Trial With Qualitative Approach
Brief Title: Sequential Practicing on Psychomotor Skill Acquisition in Undergraduate Dental Students
Acronym: Dentalpractice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nareudee Limpuangthip, DDS, PhD, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TCTR20241210005; Thai Clinical Trial.org (Other: Thai Clinical Trials Registry (TCTR))
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Undergraduate Health Professional Students; Dental Restorations; Education, Competency-Based; Dental Education and Special Care Dentistry; Dental Prosthesis
Keywords: dominant hand; sequential practice; healthcare; dental education; prosthodontic; competency

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Left: dominant - non dominant (Experimental): The left-handed participants in this arm started practicing a tooth preparation for a glass ceramic onlay using their dominant left hand during the first practicing session, followed by non-dominant right hand during the second practicing session. Each practice session is limited to 2 hours.
  Interventions: Procedure: Glass ceramic onlay preparation
- Left: non dominant (Active Comparator): The left-handed participants in this arm practicing a tooth preparation for a glass ceramic onlay using their non-dominant right hand for both the first and second practicing sessions. Each practice session is limited to 2 hours.
  Interventions: Procedure: Glass ceramic onlay preparation
- Right: dominant - non dominant (Experimental): The right-handed participants in this arm started practicing a tooth preparation for a glass ceramic onlay using their dominant right hand during the first practicing session, followed by non-dominant left hand during the second practicing session. Each practice session is limited to 2 hours.
  Interventions: Procedure: Glass ceramic onlay preparation
- Right: non dominant (Active Comparator): The right-handed participants in this arm practicing tooth preparation for glass ceramic onlay using their non-dominant left hand for both the first and second practicing sessions. Each practice session is limited to 2 hours.
  Interventions: Procedure: Glass ceramic onlay preparation

INTERVENTIONS:
Procedure: Glass ceramic onlay preparation — The participants engaged in two practice sessions, each lasting two hours. They either started with their dominant hand followed by non-dominant hand or practiced solely with their non-dominant hand. Each participant prepared a mandibular left first molar resin typodont fixed to the table for a glass ceramic onlay restoration. Preparation was conducted extraorally.

SUMMARY:
To determine the influence of hand practice sequence on psychomotor skill acquisition in a glass ceramic onlay preparation among undergraduate dental students.

DETAILED DESCRIPTION:
Effect of bilateral transfer practice on psychomotor skill acquisition among dental students remains unresolved. Bilateral transfer assumed that training one side of the body can also improve performance on the other side. Eligible participants are fourth- to sixth-year undergraduate dental students at the Faculty of Dentistry, Chulalongkorn University during the 2024 to 2025 academic year. The participants were categorized as left- or right-handed based on self-reporting. Participants enrolled two-day study with one-week separating inverval. On the first day, they learn a video presentation on glass ceramic onlay preparation followed by two practice sessions with 2-hour within each session. The practice start with either using non-dominant or dominant hand, followed by the use of non-dominant hand. One week later, they enroll two-hour practical examination on glass ceramic onlay preparation using their non-dominant hand. No practice is allowed during one-week separating interval.

ELIGIBILITY:
Inclusion Criteria:

1. The fourth- to sixth-year undergraduate dental students at a single setting of school
2. The fifth- and sixth-year students had completed laboratory and lecture courses in operative and fixed dental prosthodontics
3. The fourth-year students are enrolled in their final laboratory and lecture courses in fixed prosthodontics.

Exclusion Criteria:

Undergraduate dental students who have prior experience with onlay preparation in laboratory or clinical settings or those who are unwillingness to adhere to the study protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-07-04 (Estimated)

PRIMARY OUTCOMES:
Onlay preparation score | 3 hours
  Onlay preparation criteria using Rubic scale, assessed by the student self-assessment and one prosthodontic staff. The higher score indicates better performance of the student

SECONDARY OUTCOMES:
Qualitative measurement by focus group interview | 1 hours
  Focus group interview based on the semi-structural questionnaire regarding individual perception on the onlay preparation during practice and test sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Nareudee Limpuangthip, DDS, PhD, Principal Investigator — Chulalongkorn University

IPD SHARING:
Plan to Share IPD: No
The enrolled participants would not prefer to declare their onlay preparation score individually.